CLINICAL TRIAL: NCT04121481
Title: Clinical Study on Prodovite® VMP35 Supplement on Athletic Performance
Acronym: VMP35Sport
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Victory Nutrition International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VNI-VMP35-SPORTS-OCT 2019
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Athletic Performance
Keywords: Prodovite VMP35; RCT; Athletic Performance
MeSH Terms: interventions — Health Status; Compliance

STUDY DESIGN:
Intervention Model Description: The aim of this pilot study is to evaluate the effect of oral supplementation of Prodovite® VMP35 on exercise endurance, muscle strength, anabolic parameters and lean body mass in healthy human subjects. We hypothesize that Prodovite® VMP35 supplementation will enhance and increase exercise performance, tolerance, lean-body muscle mass, improve anabolic parameters and blood chemistry parameters in healthy human subjects. Accordingly, 150 healthy male and female subjects will be randomly assigned to receive either Prodovite® VMP35 or placebo in the form of single dose sealed containers for 90 consecutive days and muscle strength, endurance, speed, anabolic/catabolic parameters and muscle mass will be evaluated by dual energy X-ray absorptiometry (DEXA), hand-grip strength test, cycle ergometer test, spirometer assessment and assay of Blood chemistry and serum biomarkers will be evaluated before and after intervention.
Who Masked: Participant
Masking Description: Double-Blind Placebo-Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Approximately a total of 75 participants will be assigned in the Placebo Group (two divided doses will be given)
  Interventions: Dietary Supplement: Clinical Investigation on Enhanced Sports Nutrition and Performance Activities by Prodovite VMP35 Supplement; Dietary Supplement: Broad Spectrum Safety
- Treatment Group (Active Comparator): Approximately a total of 75 participants will be assigned in the Treatment Group (two divided doses will be given) Adverse Event Monitoring will be Strictly Enforced
  Interventions: Dietary Supplement: Clinical Investigation on Enhanced Sports Nutrition and Performance Activities by Prodovite VMP35 Supplement; Dietary Supplement: Broad Spectrum Safety

INTERVENTIONS:
Dietary Supplement: Clinical Investigation on Enhanced Sports Nutrition and Performance Activities by Prodovite VMP35 Supplement — Assess the Sports Nutrition efficacy of Prodovite VMP35 against the Placebo sample
  Other Names: Physical Well Being, Health Status, Detailed Lipid Profile and Blood Chemistry Analysis; Adverse Event Monitoring; Compliance
Dietary Supplement: Broad Spectrum Safety — Benefits in Sports Nutrition
  Other Names: Sports Nutrition and Health Staus

SUMMARY:
This pilot investigation will conduct a randomized placebo-controlled, double-blind study in 150 volunteers (age: 18-74 years) over a period of 90 consecutive days. A statistician will be involved in this project. Body weight, body mass index (BMI), waist circumference, blood chemistry, blood pressure and heart rate, body and hand grip strength, speed and endurance studies including open circuit spirometry-based assessment of pulmonary function will be assessed. Other parameters to be evaluated include oxygen consumption, CO2 production and metabolic parameters, VO2 max, respiratory exchange ratio (RER), anaerobic threshold, ventilatory equivalents for oxygen (VE/V02) and exhaled carbon dioxide (VE/VC02)2,3. Subjects will participate in completed maximal graded exercise tests (GXT) on a treadmill or in set distance open-field sprints using open-circuit spirometry. Lower and Upper Body Strength will be evaluated. E-Diary will be provided to all participants. Survey Monkey program will be provided to all subjects and regularly updated by all study participants daily and endorsed by the co-Principal Investigator.

DETAILED DESCRIPTION:
A novel patented Prodovite® VMP35 Multi-Nutrient-Complex (MNC), a vitamin, mineral, and phytonutrient encapsulated liquid formulation, was prepared using a novel proprietary SK713 SLP multi-lamellar clustoidal non-GMO phospholipid Prodosome nutrient absorption/delivery technology in a state-of-the-art multistep cGMP and NSF-certified manufacturing facility. This developmental technology is biodegradable and biocompatible. Preliminary study in our laboratory demonstrated the efficacy of Prodovite® VMP35 in Sports Nutrition. We hypothesize that Prodovite® VMP35 supplement will enhance athletic performance, lean-body muscle mass, increase exercise tolerance, and improve anabolic parameters in healthy human subjects. The aim of this pilot study is to evaluate the effect of oral supplementation of Prodovite® VMP35 on exercise endurance, muscle strength, anabolic parameters and lean body mass in healthy human subjects. We hypothesize that Prodovite® VMP35 supplementation will enhance and increase exercise performance, tolerance, lean-body muscle mass, improve anabolic parameters and blood chemistry parameters in healthy human subjects. Accordingly, 150 healthy male and female subjects will be randomly assigned to receive either Prodovite® VMP35 or placebo in the form of single dose sealed containers for 90 consecutive days and muscle strength, endurance, speed, anabolic/catabolic parameters and muscle mass will be evaluated by dual energy X-ray absorptiometry (DEXA), hand-grip strength test, cycle ergometer test, spirometer assessment and assay of Blood chemistry and serum biomarkers will be evaluated before and after intervention.

ELIGIBILITY:
Inclusion and Exclusion Criteria

Inclusion criteria

1. Agrees to written as well as audio-visual informed consent
2. Ability to understand the risks/benefits of the study protocol
3. Healthy male and female, human subjects 18-74 years of age
4. Subjects experienced with at least six months of regular athletic performance training

AND

Exclusion criteria

1. Uncooperative Subjects
2. Subjects with chronic illness (diabetes, cardiovascular disease, cancer, arthritis, etc) or those on prescription medication excluded (except for birth control pills)
3. Any conditions that prevent the subject from participating in physical activities.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Anthropometric Measurements: Body Weight | Over a Period of 90-Consecutive Days
  Body Weight (Kilograms)
Anthropometric Measurements: Height | Over a Period of 90-Consecutive Days
  Height (Meters)
Anthropometric Measurements: Waist Circumference | Over a Period of 90-Consecutive Days
  Waist Circumference (Meters)
Anthropometric Measurements: Waist-Hip Ratio | Over a Period of 90-Consecutive Days
  Waist : Hip Ratio
Anthropometric Measurements: Blood Pressure (mmHg) | Over a Period of 90-Consecutive Days
  Blood Pressure (mmHg)
Body Composition and Bone Mineral Density: DEXA (GE) | Over a Period of 90-Consecutive Days
  DEXA and Bone Mineral Density
Ergometric Assessment: Treadmill | Over a Period of 90-Consecutive Days
  Ergometric measurements
Handgrip Dynamometer | Over a Period of 90-Consecutive Days
  Handgrip strength
Respiration Quality and Rate: Spirometer | Over a Period of 90-Consecutive Days
  Respiration Quality, VO2 and VCO2 assessments
Endurance Studies | Over a Period of 90 Consecutive Days
  Cycle Ergometer, Bench Press and Leg Press

SECONDARY OUTCOMES:
Lipid Profile | Over a Period of 90-Consecutive Days
  Complete Lipid Profile
Total Blood Chemistry | Over a Period of 90-Consecutive Days
  Blood Chemistry

CONTACTS AND LOCATIONS:
Overall Officials: BRUCE S MORRISON, DO, Principal Investigator — SPORTS NUTRITION & FAMILY MEDICINE
Locations (1):
- Champions Sports Performance & Hardcore Serious Fitness, Cornelius, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IT IS A RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND STUDY

REFERENCES:
- [Result] Corbier JR, Downs BW, Kushner S, Aloisio T, Bagchi D, Bagchi M. VMP35 MNC, a novel iron-free supplement, enhances cytoprotection against anemia in human subjects: a novel hypothesis. Food Nutr Res. 2019 May 9;63. doi: 10.29219/fnr.v63.3410. eCollection 2019. PMID 31105509